CLINICAL TRIAL: NCT05551754
Title: Acute Effects of Ketone Supplementation on Subjective and Objective Responses to Alcohol in Healthy Volunteers
Brief Title: Acute Effects of Ketone Supplement on Responses to Alcohol Challenge in Healthy Volunteers
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 852002
Record Dates: First submitted 2022-09-15; First posted 2022-09-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Drinking
Keywords: Ketone Ester
MeSH Terms: conditions — Alcohol Drinking | interventions — 1,3-butylene glycol; Ethanol

STUDY DESIGN:
Intervention Model Description: Placebo controlled, randomized, crossover trial in 10 healthy volunteers
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ketone supplement (Active Comparator): Subjects will drink single dose of ketone supplement 25g
  Interventions: Dietary Supplement: Ketone Supplement; Other: Alcohol Beverage
- Placebo beverage (Placebo Comparator): Subjects will drink single dose of placebo beverage that will look and taste the same as ketone supplement.
  Interventions: Other: Alcohol Beverage

INTERVENTIONS:
Dietary Supplement: Ketone Supplement — Drink a single dose of ketone supplement 25g
  Other Names: ketone supplement, D-hydroxybutyric acid and 1,3 butanediol
  Arms: ketone supplement
Other: Alcohol Beverage — Subjects will drink about 2 ½ standard alcohol beverages, based on their weight to reach a breath alcohol level of 0.050%

SUMMARY:
This is a single blinded, randomized trial to evaluate the immediate subjective and objective effects of alcohol after a dose ketone supplement compared to a placebo in 10 health volunteers. Subjects will complete 2 lab visits where they consume a dose of alcohol (based on weight), to bring their breath alcohol concentration to about 0.050%. Participants will randomly receive ketone supplement at one lab and the placebo at the next lab.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the immediate subjective and objective effects of alcohol after consuming a ketone supplement beverage, compared to a placebo beverage (an inactive substance). Participants will not know which lab they receive the ketone drink, however they will be asked to drink an alcohol beverage (based on weight), to bring breath alcohol concentration (BrAC) to about 0.050% at each lab visit.

The goal of the study is to see how measure subjective effects of alcohol, once after drinking the ketone supplement and once after drinking a placebo beverage. The study will use questionnaires, blood, and breath alcohol tests to see how subjects body and brain experience alcohol. The study is also interested in if the ketone supplement makes people want to drink alcohol more or less.

Consent and Screening Session (approximately 3 hrs)

The following will occur at the screening session, following signed consent:

* First, subjects will be asked to show a legal photo ID and then undergo a breathalyzer test to ensure that they are able to make a well-reasoned decision about whether or not to participate in the study. The BrAC must be at 0.000% to complete this visit.
* Demographic information, such as date of birth, age, biological sex, marital status, education, race, and ethnicity will be collected.
* Subjects will be asked to provide current information about address and contact information to register them as a patient at the University of Pennsylvania, if they have not been a patient here before.
* Approximately 2 tablespoons of blood for standard laboratory tests will be drawn. It is possible that bloodwork will need to be repeated due to unforeseen events (abnormal findings or potential lab errors).
* Subject's will be asked to provide a urine sample for routine urinalysis, drug screen, and a pregnancy test in women who are able to become pregnant.
* Study personnel will measure vital signs (blood pressure and pulse), weight, and height. Subject's will be asked to complete a questionnaire about current and past medical history and any medications currently taking.
* Study personnel will complete a brief psychiatric interview and ask about alcohol and cigarette use over the past 90 days.

Staff will confirm eligible within 5 business days after the screening visit, to schedule the rest of the study visits.

Lab visits (approximately 5 1/2 hrs) The following will occur on the day of the two lab visits as a participant.

* Subject's are asked to not eat or drink anything except water after midnight the day before and on the day of the lab visit. A light meal will be provided on the lab days, after staff takes a BrAC (must be 0.000% to continue), preforms a finger stick for blood glucose level (must be below 140), measures weight, and vital signs.
* Subjects will be asked to provide a urine sample to conduct a drug screen, and a pregnancy test (for woman able to become pregnant).
* Staff will review the current list medications and vitamins provided at the screening visit and ask if anything has changed?
* Subjects will be asked about alcohol and drug use history since the last visit.
* Approximately 1 hour after the light meal, subjects will be asked to drink the ketone supplement or placebo beverage.
* Approximately 30 minutes after drinking the beverage, subjects will be asked to drink an alcohol beverage based on weight in 15 minutes. Staff will record the BrAC, draw blood and ask subjects to complete questionnaire as listed in the below table.
* Staff will ask about any side effects that may occur throughout the lab procedures.
* During the lab day between study procedures, subjects may read books, magazines, or watch videos.
* After a snack, staff will check the final BrAC and ask again about any side effects. The second visit will be scheduled at least 2 days after the first visit and will follow the same procedures. Subjects may leave with a BrAC below 0.010.

Table of assessments on Lab Visits:

* Approximate study times • Procedure
* 10:30am • BrAC1, vital signs, urine sample
* 10:40am • light meal
* 11:00am • Review of medications currently taking, and review of alcohol and drug use since last visit
* 12:00pm • Ketone supplement or placebo drink
* 12:20pm • BrAC 2, and 3 questionnaires
* 12:30pm • Finger stick
* Alcohol administration
* 12:45pm • BrAC 3, and blood draw 1
* 1:00pm • BrAC 4, and 2 questionnaires
* 1:15pm • BrAC 5, and blood draw 2
* 1:30pm • BrAC 6, and 2 questionnaires
* 2:00pm • BrAC 7, Blood draw 3, and 3 questionnaires
* 2:30pm • BrAC 8
* 3:00pm • BrAC 9
* 3:30pm • BrAC 10, blood draw 4, and 3 questionnaires
* 3:50pm • Snack
* 4:00pm • Final BrAC end of visit.

Follow-up Visit (approximately 5 minutes): A follow-up phone call will occur the day after each lab visit and the following will occur:

• Staff will ask about any side effects that may have been experienced.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide signed, informed consent and commit to completing the alcohol lab studies.
2. All subjects must report at least one occasion in the prior month of drinking at least 2 drinks on a single day.

Exclusion Criteria:

1. Unwilling or unable to refrain from use, within 24 hours of alcohol lab procedures, psychoactive medications or medications that may affect study results.
2. Current DSM-5 diagnosis of a major psychiatric disorder (other than nicotine use disorders, or marijuana use disorders) (identified by clinical examination or the structured interview) that could interfere with study participation or make it hazardous for the subject.
3. Currently taking a medication that could interfere with study participation or make it hazardous for the subject to participate. (e.g., anticholinergics; antipsychotics; lithium; psychotropic drugs not otherwise specified)
4. Positive urine drug screen positive for all substances but marijuana on study visits (may be repeated once and if the result is negative on repeat it is not exclusionary).
5. A baseline breath alcohol concentration of greater than 0.00% on study visit prior to alcohol tolerance test
6. A current, clinically significant physical disease or abnormality on the basis of medical history, or routine laboratory evaluation that can impact brain function, the use of a ketone supplement or the use of alcohol (e.g., epilepsy, diabetes, irritable bowel syndrome, Crohn's disease, liver disease, kidney disease, kidney stones, chronic metabolic acidosis or a cardiomyopathy as determined by history and clinical exam).
7. Currently suffering from or with a history of stroke and/or stroke related spasticity.
8. Head trauma with loss of consciousness for more than 30 minutes or associated with skull fracture or inter-cranial bleeding or abnormal MRI. (self-report, medical history).
9. Weight greater than 225lbs (Need to cap amount of alcohol give based on weight to individuals).
10. Judged by the principal investigator or his designee to be an unsuitable candidate for study participation.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Acute effects of breath/blood alcohol levels in response to ketone supplement verse placebo | 4 hours
  Change in breath/blood alcohol levels (grams per 210 Liters of breath) in response to ketone supplement verse placebo

SECONDARY OUTCOMES:
Acute effects of subjective reports of intoxication and alcohol craving in response to ketone supplement verse placebo after alcohol drinks. | 4 hours
  Change in subjective effects are measured using the Drug Effects Questionnaire (DEQ): A 5-item scale assessing the extent to which participants (1) feel any DRUG EFFECTS, (2) feel HIGH, (3) LIKE the effects, (4) DISLIKE the effects, and (5) want MORE of the substance using a 100-mm visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Corinde Wiers, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Studies of Addiction, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No